CLINICAL TRIAL: NCT02197663
Title: Clinical Evaluation of Acupuncture on the Complications of Cerebral Vascular Accident
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: the numbers of drop-out patients are more than we anticipate
Sponsor: China Medical University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CMUH102-REC2-015
Record Dates: First submitted 2014-06-08; First posted 2014-07-23 (Estimated); Last update posted 2015-10-22 (Estimated); Status verified 2015-10

CONDITIONS: Stroke
Keywords: acupuncture; stroke; Randomized Controlled Trial
MeSH Terms: conditions — Stroke | interventions — Acupuncture Therapy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Acupuncture (Experimental): The total course of the acupuncture contains 24times(about 3 months). The acupoints are fixed and located over head and limbs.
  Interventions: Procedure: acupuncture(44mm in length and 32-gauge)
- sham acupuncture (Sham Comparator): The total course of the acupuncture contains 24times(about 3 months). The acupoints are fixed and 1cm away from meridian and no acupoints over head were chosen.
  Interventions: Procedure: acupuncture(44mm in length and 32-gauge)

INTERVENTIONS:
Procedure: acupuncture(44mm in length and 32-gauge) — The whole course of the acupuncture contains 24times(about 3 months). The acupoints are fixed and located over head and limbs.
  The whole course of the sham acupuncture contains 24times(about 3 months). The acupoints are fixed and 1cm away from meridian and no acupoints over head were chosen.
  Other Names: acupuncture(4.4cm in length and 32-gauge); shame acupuncture(1.27 cm in length and 40-gauge)

SUMMARY:
The lifestyle of Taiwanese people has been changed over the past decade with the improvement of economic growth, environmental sanitation and the quality of medical care. Now the investigators pay more attention to the increasing risk of people's diseases of civilization than people's malnutrition and poor quality of environmental sanitation. The cerebrovascular accident (CVA) leads to death and bio-psycho-social dysfunction. The medical care of the patient of cerebrovascular accident cause a lot of money and is a burden of our country.

Our study emphasizes that acupuncture change bio-psycho-social aspects of the patient with cerebrovascular accident. The investigators use some scales to assess efficacy of acupuncture, such as Barthel index, National Institute of Health Stroke Scale, Visual Analogue Scale, Instrumental Activities of Daily Living and Hamilton Depression Rating Scale.

Besides, the investigators notice that there are few journals about acupuncture effect of treating depression following cerebral vascular accident. The investigators may underestimate the amount of people having post-stroke depression. So the investigators use Hamilton Depression Rating Scale to Assess the post-stroke depression of cerebral vascular accident patient.

By assessing bio-psycho-social level of CVA patient, the investigators hope this study will offer them more "Holistic Health Care".

DETAILED DESCRIPTION:
We want to assess the effect of acupuncture on stroke patients. The study is a double-blind randomized controlled trial. We need 80 patients altogether. The Inclusion Criteria:

(1)first time stroke(ischemic or hemorrhagic stroke) with paresis or plegia

Exclusion Criteria:

(1)transient ischemic attack (2)brain tumor, brain trauma (3)recurrent stroke (4)multiple organs failure, cancer The whole course of the acupuncture contains 24times(about 3 months). The acupoints are fixed and located over head and limbs.

The whole course of the sham acupuncture contains 24times(about 3 months). The acupoints are fixed and 1cm away from meridian and no acupoints over head were chosen.

The investigators use Barthel index, National Institute of Health Stroke Scale, Hamilton Depression Rating Scale, Instrumental activities of daily living scale and Visual Analogue Scale to assess the effect of acupuncture on stroke patients. Four times of assessment are as below: baseline, after 8th treatment, after 16th treatment, after 24th treatment (the last time of treatment). The course of treatment should be completed within 3 months.

ELIGIBILITY:
Inclusion Criteria:

* first time stroke(ischemic or hemorrhagic stroke) with paresis or plegia

Exclusion Criteria:

* transient ischemic attack
* brain tumor, brain trauma
* recurrent stroke
* multiple organs failure, cancer

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2013-04; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Change from baseline in Barthel index at 8 weeks | Baseline and 8 weeks
Change from baseline in Barthel Index at 16 weeks | Baseline, 16 weeks
Change from baseline in Barthel Index at 24 weeks | Baseline, 24 weeks
Change from baseline in National Institute of Health Stroke Scale at 8 weeks | Baseline, 8 weeks
Change from baseline in National Institute of Health Stroke Scale at 16 weeks | Baseline, 16 weeks
Change from baseline in National Institute of Health Stroke Scale at 24 weeks | Baseline, 24 weeks
Change from baseline in Instrumental Activities of Daily Living Scale at 8 weeks | Baseline, 8 weeks
Change from baseline in Instrumental Activities of Daily Living Scale at 16 weeks | Baseline, 16 weeks
Change from baseline in Instrumental Activities of Daily Living Scale at 24 weeks | Baseline, 24 weeks
Change from baseline in Hamilton Depression Rating Scale at 8 weeks | Baseline, 8 weeks
Change from baseline in Hamilton Depression Rating Scale at 16 weeks | Baseline,16 weeks
Change from baseline in Hamilton Depression Rating Scale at 24 weeks | Baseline, 24 weeks

SECONDARY OUTCOMES:
Change from baseline in Visual Analogue Scale at 8 weeks | Baseline, 8 weeks
Change from baseline in Visual Analogue Scale at 16 weeks | Baseline,16 weeks
Change from baseline in Visual Analogue Scale at 24 weeks | Baseline, 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Yu-Chen Lee, PHD, Study Director — Department of Acupuncture, China Medical University Hospital
Locations (1):
- Department of Acupuncture, China Medical University Hospital, Taichung, Taiwan